CLINICAL TRIAL: NCT02316886
Title: a Multinational, Multicenter, Prospective, Open-label, Active-treatment-controlled Randomized Trial: Preventive PCI or Medical Therapy Alone for Vulnerable Atherosclerotic Coronary Plaque_PREVENT Trial
Brief Title: Preventive PCI or Medical Therapy Alone for Vulnerable Atherosclerotic Coronary Plaque
Acronym: PREVENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2014-13
Record Dates: First submitted 2014-12-01; First posted 2014-12-15 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease; Plaque, Atherosclerotic
Keywords: coronary intervention; Vulnerable Plaque; Insignificant Stenosis; Bioresorbable Vascular Scaffold; Everolimus Eluting stent
MeSH Terms: conditions — Coronary Artery Disease; Plaque, Atherosclerotic | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coronary intervention (Experimental): bioabsorbable vascular scaffolds (BVS) (early period) or everolimus-eluting stents (middle and late period) +Optimal Medical Treatment
  Interventions: Device: Coronary intervention
- Optimal Medical Treatment (Active Comparator): Optimal Medical Treatment
  Interventions: Drug: Optimal Medical treatment

INTERVENTIONS:
Device: Coronary intervention — bioabsorbable vascular scaffolds (BVS) (early period) or everolimus-eluting stents (middle and late period) + Optimal Medical Treatment
  Arms: Coronary intervention
Drug: Optimal Medical treatment
  Arms: Optimal Medical Treatment

SUMMARY:
The primary aim of the trial is to determine whether preventive PCI with bioabsorbable vascular scaffolds (BVS) (early period) or everolimus-eluting stents (middle and late period) plus optimal medical therapy (OMT) on functionally insignificant (FFR > 0.80) vulnerable coronary plaque, as determined by intracoronary imaging, would result in a significant reduction of the primary composite outcome of death from cardiac causes, target-vessel myocardial infarction (MI), target-vessel revascularization (TVR), and hospitalization for unstable or progressive angina at 2 years, when compared with OMT alone.

DETAILED DESCRIPTION:
Sub-analysis for each imaging test will be performed as below;

* NIRS(Near-infrared spectroscopy)
* OCT(Optical coherence tomography)
* VH-IVUS(IVUS-derived virtual histology)
* IVUS(Intravascular ultrasonography)

Extended follow-up:

Considering the nature of functionally insignificant coronary stenosis with vulnerable plaque, most subjects are watched for extended follow-up after the planned 2-year follow-up time point.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Patients with suspected or known Coronary artery disease who are undergoing invasive cardiac catheterization
* Patients with at least one significant stenosis (diameter stenosis >50%) with Fractional Flow Reserve (FFR) >0.80 and meeting two of the following criteria:

  1. MLA(minimal luminal area)<4mm2
  2. Plaque burden>70%
  3. Large lipid-rich plaque on NIRS(Intracoronary Near-Infrared Spectroscopy), defined as MaxLCBI4mm>315
  4. TCFA(thin-cap fibroatheroma) defined as fibrous cap thickness <65 μm and arc >90° on optical coherence tomography (OCT) or ≥10% confluent necrotic core with >30° abutting the lumen in three consecutive slices on Virtual-histology intravascular ultrasound (VH-IVUS)
* Eligible for percutaneous coronary intervention with Absorb Bioresorbable Vascular Scaffold or Everolimus Eluting Stent
* Reference vessel diameter 2.75-4.0
* Lesion length ≤ 40mm
* Willing and able to provide informed written consent

Exclusion Criteria:

* Patients for whom the preferred treatment is CABG(Coronary artery bypass grafting)
* Patients with stented lesions
* Patients with bypass graft lesions
* Patients with three or more target lesions
* Patients with two target lesions in the same coronary territory
* Patients with heavily calcified or angulated lesions
* Patients with bifurcation lesions requiring 2 stenting technique
* Patients with contraindications to or planned discontinuation of dual antiplatelet therapy within 1 year
* Patients with life expectancy <2 years
* Patients with planned cardiac or major noncardiac surgery
* Woman who are breastfeeding, pregnant or planning to become pregnant during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1608 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Target vessel failure | 2 years
  target-vessel failure, which was defined a composite of death from cardiac causes, target-vessel myocardial infarction, ischemic-driven target-vessel revascularization, or hospitalization for unstable or progressive angina

SECONDARY OUTCOMES:
Death from cardiac causes | 2 years
Target-vessel myocardial infarction | 2 years
Ischemic-driven target-vessel revascularization | 2 years
Hospitalization for unstable or progressive angina | 2 years
Death from all, cardiac, or noncardiac causes | 2 years
Myocardial infarction | 2 years
  Periprocedural or spontaneous, target-vessel or non-target-vessel related
Repeat revascularization | 2 years
  Repeat revascularization (target-vessel or non-target-vessel, ischemia-driven or non-ischemia-driven)
Any hospitalization for cardiac or noncardiac causes | 2 years
Target-lesion failure | 2 years
  cardiac death, target-vessel myocardial infarction or ischemia-driven target-lesion revascularization
Major adverse cardiac event | 2 years
  defined as death from cardiovascular causes, nonfatal myocardial infarction, or unplanned rehospitalization due to unstable or progressive angina
Composite of any death, myocardial infarction, or repeat revascularization | 2 years
  A composite endpoint is an endpoint that is a combination of multiple clinical endpoints. An event is considered to have occurred if any one of several different events is observed.
Rate of Scaffold or stent thrombosis | 2 years
Rate of Stroke | 2 years
Rate of Bleeding events | 2 years
  life-threatening or disabling, major or minor
Rate of Nonurgent revascularization procedures | 2 years
Functional class | 2 years
  It is assessed by the Canadian Cardiovascular Society (CCS) Classification at each point in time.
  The Canadian Cardiovascular Society (CCS) classification has four categories; the minimum and maximum values are 1 and 4 respectively. A higher score means a worse outcome.
Number of anti-anginal medications administered | 2 years
  Number of anti-anginal medication at each point in time

CONTACTS AND LOCATIONS:
Overall Officials: Duk-woo Park, MD, Principal Investigator — Asan Medical Center
Locations (18):
- Columbia University Medical Center, New York, New York, United States
- Kyoto University Hospital, Kyoto, Japan
- Christchurch Hospital and Canterbury DHB, University of Otago, Christchurch, New Zealand
- South Korea (14):
  - Asan Medical Center, Seoul, Songpa-gu
  - Hallym University Sacred Heart Hospital, Anyang
  - Gangwon National Univ. Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Hospital, Incheon
  - ChonBuk National University Hospital, Jeonju
  - Samsung Medical Center, Seoul
  - Seoul National University hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Bundang Cha Medical Center, Sŏngnam
  - Seoul National University Bundang hospital, Sŏngnam
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park SJ, Ahn JM, Kang DY, Yun SC, Ahn YK, Kim WJ, Nam CW, Jeong JO, Chae IH, Shiomi H, Kao HL, Hahn JY, Her SH, Lee BK, Ahn TH, Chang KY, Chae JK, Smyth D, Mintz GS, Stone GW, Park DW; PREVENT Investigators. Preventive percutaneous coronary intervention versus optimal medical therapy alone for the treatment of vulnerable atherosclerotic coronary plaques (PREVENT): a multicentre, open-label, randomised controlled trial. Lancet. 2024 May 4;403(10438):1753-1765. doi: 10.1016/S0140-6736(24)00413-6. Epub 2024 Apr 8. PMID 38604213
- [Derived] Ahn JM, Kang DY, Lee PH, Ahn YK, Kim WJ, Nam CW, Jeong JO, Chae IH, Shiomi H, Kao PHL, Hahn JY, Her SH, Lee BK, Ahn TH, Chang K, Chae JK, Smyth D, Stone GW, Park DW, Park SJ; PREVENT Investigators. Preventive PCI or medical therapy alone for vulnerable atherosclerotic coronary plaque: Rationale and design of the randomized, controlled PREVENT trial. Am Heart J. 2023 Oct;264:83-96. doi: 10.1016/j.ahj.2023.05.017. Epub 2023 Jun 2. PMID 37271356